CLINICAL TRIAL: NCT06185075
Title: Influence of Implant Crown Transmucosal Contour Design on Soft and Hard Tissue Clinical Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Muhammad Saleh, Clinical Assistant Professor, Periodontics and Oral Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00208140 Substudy
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gum Disease
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Straight transmucosal contour (Active Comparator): Implant crown will be designed with a straight transmucosal contour
  Interventions: Procedure: Implant crown delivery
- Concave transmucosal contour (Active Comparator): Implant crown will be designed with a concave transmucosal contour
  Interventions: Procedure: Implant crown delivery

INTERVENTIONS:
Procedure: Implant crown delivery — Dental implant crown will be designed, fabricated by a dental lab, and delivered.

SUMMARY:
This study will evaluate how the crown's shape under the gums will influence the gum tissue around dental implants.

DETAILED DESCRIPTION:
This research is studying the transmucosal contour, or shape of crowns (white-colored tooth structure that sits above the gum) under the gums on dental implants. Participants will be randomly selected for the dental implant crown to be designed with either a straight or concave transmucosal contour, and followed up on for 1 year after crown delivery.

ELIGIBILITY:
Inclusion criteria

* Be a current participant of HUM00208140 main study
* Have a dental implant that is ready to be restored (placed at least 3 months ago and healing is adequate)

Exclusion Criteria:

• The dental implant crown was already delivered.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss around dental implant | 6 months and 12 months after crown delivery
  Measured from radiographs in mm
Gum tissue thickness | 6 months and 12 months after crown delivery
  Measured from intraoral scan in mm
Gingival margin height | 6 months and 12 months after crown delivery
  Measured from intraoral scan in mm
Amount of keratinized gingiva | 6 months and 12 months after crown delivery
  Measured clinically in mm

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleh, BDS, MSD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No